CLINICAL TRIAL: NCT00207168
Title: A Randomized, Multi-center, Open Label Study in Well Controlled Treatment-experienced HIV- Infected Patients to Assess Compliance With a Once-daily Regimen
Brief Title: To Assess Compliance With a Once-daily Regimen of Lamivudine, Efavirenz and Didanosine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry); Dohme Australia (Unknown)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI454-194; The TEddI Study
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-04

CONDITIONS: AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Compliance

INTERVENTIONS:
Behavioral: Compliance

SUMMARY:
To assess compliance of once daily dosing to assess their benefits in terms of potency and safety as well as their impact on adherence and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older, required lab results, currently taking no more than two of the proposed once daily arm medications with medications administered twice daily and women of child bearing potential.

Exclusion Criteria:

* virological failure, serious medical condition, known toxicities to any of the once daily arm medications, lab abnormalities, women who are pregnant/breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2004-04; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To determine over 24 weeks the levels of adherence in two groups of HIV-infected subjects randomized to receive either a once daily 3-drug regimen or to continue a minimum 3-drug regimen requiring more frequent dosing.

SECONDARY OUTCOMES:
To demonstrate that once daily therapy is not-inferioir to continued multiple dosing in terms of proportion of patients with treatment failure.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb